CLINICAL TRIAL: NCT06473610
Title: Residual Embolism Evaluated With Single Photon Emission Computed Tomography - The RESPECT Cohort
Brief Title: Residual Embolism Evaluated With Single Photon Emission Computed Tomography
Acronym: RESPECT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 23CH190; 2024-A00613-44 (Other: ANSM)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Circulation Obstruction
Keywords: scintigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Major progress achieved in diagnostic and therapeutic strategies has substantially improved the short-term prognosis of patients with pulmonary embolism (PE). These improvements have led to a shift from an acute to a chronic condition of venous thromboembolism, justifying the recent development of Chronic Thrombo-embolic Disease (CTED). In most of the situations, it is due to a residual pulmonary vascular obstruction (RPVO) which can be assessed by pulmonary scintigraphy.

DETAILED DESCRIPTION:
Planar ventilation/perfusion (V/Q) scintigraphy is the gold standard, but for several months, V/Q single photon emission computed tomography (SPECT) is recommended in the guidelines.

The aim of this study is to evaluate the performances of various SPECT protocols to quantified RPVO and compared to planar scintigraphy to evaluate the RPVO.

ELIGIBILITY:
Inclusion Criteria:

* Patient addressed to nuclear medicine department of Saint-Etienne public hospital for V/Q pulmonary SPECT-CT assess to rule out perfusion obstruction, admitted for a suspicion of pulmonary hypertension (PH), or a persistent dyspnea after PE
* Patient affiliated ou beneficiary of social security.

Exclusion Criteria:

* Pregnant patient.
* Patient addressed to nuclear medicine department for acute pulmonary embolism.
* Impossibility of the entire protocol acquisitions realization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with V/Q pulmonary SPECT-CT assess to rule out perfusion obstruction, patients admitted for a suspicion of PH, or a persistent dyspnea after PE
Sampling Method: Non-Probability Sample
Enrollment: 358 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
RPVO (%) | At inclusion
  Evaluation of the RPVO establish with Meyer score (planar scintigraphy, 2D). The higher the percentage, the greater the obstruction of the lung
Segmental visual score | At inclusion
  Evaluation of segmental visual score (SPECT-CT , 3D) The higher the percentage, the greater the obstruction of the lung

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Benoit BONNEFOY, MD, Principal Investigator — CENTRE HOSPITALIER DE SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No